CLINICAL TRIAL: NCT03012997
Title: Effects of Hyperoxia on Oxidative Stress in Patients Undergoing Open Heart Surgery
Brief Title: Effects of Hyperoxia on Open Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Collaborators: Koşuyolu Kartal Heart Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Guniz M.Koksal, Professor Anesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: KK01
Record Dates: First submitted 2016-12-09; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Heart Valve Disease; Coronary (Artery) Disease
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Comparator: 40% oxygen (Active Comparator): Patients in this group will be ventilated with fraction of inspired oxygen 40% during the induction, surgery and in Postoperative care unit.
  Interventions: Other: Fraction of inspired oxygen 40%
- Active Comparator: 100% oxygen (Active Comparator): Patients in this group will be ventilated with fraction of inspired oxygen during 100% induction and with 60-70% ( determined according to the arterial blood gas sample results) during surgery and in Postoperative care unit.
  Interventions: Other: Fraction of inspired oxygen 100%

INTERVENTIONS:
Other: Fraction of inspired oxygen 40%
  Arms: Active Comparator: 40% oxygen
Other: Fraction of inspired oxygen 100%
  Arms: Active Comparator: 100% oxygen

SUMMARY:
Patients undergoing Open Cardiac Surgery will be randomized into two groups. Group I will be ventilated with 40% Fio2 during induction, surgery and in Postoperative care unit. Group II will be ventilated with 100% Fio2 during induction and with 60-70% ( determined according to the arterial blood gas sample results) during surgery and in Postoperative care unit.

Hemodynamic parameters ( systolic arterial pressure, diastolic arterial pressure, heart rate ), Arterial blood gas samples ( PaO2, PaCO2, pH, Oxygen saturation, Lactate), and pre and post cardiopulmonary bypass Superoxide dismutase and malonyl aldehyde levels.

ELIGIBILITY:
Inclusion Criteria:

* ASA II-III
* Patients with EF higher than 50%.
* patients undergoing elective open heart surgery on pump ( CABG, Valve Replacement)

Exclusion Criteria:

* patients with Diabetes Mellitus
* patients with COPD
* Patients with Cerebral Vascular Disease
* Patients with hypoxia in Arterial blood gas samples ( PaO2 lower than 80 mmHg) and hypercarbia (PaCO2 higher than 45 mmHg)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
change in Malondialdehyde (MDA) (nmol/mg pr) levels (as a biomarker for oxidative stress ) and Superoxide dismutase (SOD) (nmol/mg pr) levels as a biomarker for antioxidant response in the plasma between "before" and "after" cardiopulmonary bypass | 72 hours
  As primary outcome, the effects of different inspired oxygen fractions on oxidative stress and anti-oxidant response in before and after cardiopulmonary bypass will be evaluated

SECONDARY OUTCOMES:
Partial pressure of oxygen(mmHg), | 72 hours
  Partial pressure of oxygen(mmHg) in arterial-blood-gas samples before induction, following induction, before and after cardiopulmonary bypass, before extubation and following extubation, postoperative 24 and 72th hours.
Partial pressure of carbondioxide(mm Hg) | 72 hours
  ,Partial pressure of carbondioxide(mm Hg) in arterial-blood-gas samples before induction, following induction, before and after cardiopulmonary bypass, before extubation and following extubation, postoperative 24 and 72th hours.
lactate (mmol/l) | 72 hours
  lactate (mmol/l) levels in arterial blood gas samples before induction, following induction, before and after cardiopulmonary bypass, before extubation and following extubation, postoperative 24 and 72th hours.
ph values | 72 hours
  ph values in arterial blood gas samples before induction, following induction, before and after cardiopulmonary bypass, before extubation and following extubation, postoperative 24 and 72th hours.
systolic arterial pressure (mmHg), | 72 hours
  systolic arterial pressure (mmHg), levels before induction, following induction, before and after cardiopulmonary bypass, before extubation and following extubation, postoperative 24 and 72th hours.
diastolic arterial pressure (mmHg) | 72 hours
  diastolic arterial pressure (mmHg) levels before induction, following induction, before and after cardiopulmonary bypass, before extubation and following extubation, postoperative 24 and 72th hours.
Oxygen saturation (%) | 72 hours
  Oxygen saturation (%) levels in arterial blood gas samples before induction, following induction, before and after cardiopulmonary bypass, before extubation and following extubation, postoperative 24 and 72th hours.
heart rate (beat/min) | 72 hours
  heart rate (beat/min) levels before induction, following induction, before and after cardiopulmonary bypass, before extubation and following extubation, postoperative 24 and 72th hours.

CONTACTS AND LOCATIONS:
Overall Officials: Guniz Koksal, Professor, Study Director — Istanbul University
Locations (2):
- Turkey (Türkiye) (2):
  - Kartal Kosuyolu Training and Research Hospital, Istanbul, Marmara
  - Kartal Kosuyolu Training and Research Hospital, Istanbul

REFERENCES:
- [Background] Koksal GM, Dikmen Y, Erbabacan E, Aydin S, Cakatay U, Sitar ME, Altindas F. Hyperoxic oxidative stress during abdominal surgery: a randomized trial. J Anesth. 2016 Aug;30(4):610-9. doi: 10.1007/s00540-016-2164-7. Epub 2016 Mar 21. PMID 27001081